CLINICAL TRIAL: NCT03245463
Title: Evaluation of Different Methods of Teaching Self-management Strategies to Patients With Symptomatic Knee Osteoarthritis
Brief Title: Evaluation of Methods of Teaching Self-management Strategies to Patients With Symptomatic Knee Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2017-0731
Record Dates: First submitted 2017-08-07; First posted 2017-08-10 (Actual); Results first posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-10

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Teaching Method A (Active Comparator): Patient will receive an educational handout on self-management strategies. Patient will be asked to take the handout home to read and to call the office if he/she has any questions.
  Interventions: Other: Educational handout; Drug: Hyaluronic Acid
- Teaching Method B (Active Comparator): Patient will receive an educational handout on self-management strategies. A provider will review the handout with the patient (approximately 5 minutes including a question-and-answer session).
  Interventions: Other: Educational handout; Other: Verbal script; Drug: Hyaluronic Acid

INTERVENTIONS:
Other: Educational handout — The educational handout will include information on self-management strategies.
Other: Verbal script — The verbal script will include details on self-management strategies that will be reviewed with the patient.
  Arms: Teaching Method B
Drug: Hyaluronic Acid — All study patients are undergoing injections with hyaluronic acid prior to the administration of the teaching method. The injections are standard of care and are required as part of the inclusion criteria.

SUMMARY:
Symptomatic knee osteoarthritis greatly impacts the quality of life, mobility, independence, and even safety of the individuals who suffer from it. One of the most powerful tools for these patients can be education on self-care and self-management strategies that can be taught to a patient by a physician, physical or occupational therapist, or a nurse. These self-management strategies can help patients treat daily stiffness through exercise or manage flares of osteoarthritis. There is a lack of consensus on the best teaching methods to accomplish the goal of educating our patients. Feedback from both patients and providers regarding teaching methods is needed. This study will evaluate teaching methods on self-management strategies for patients who are undergoing hyaluronic acid injections for knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patients of co-investigator physicians
* Age 18+ years
* Diagnosis of symptomatic knee osteoarthritis
* Scheduled for a hyaluronic acid injection into the knee
* Provider is available to administer teaching method

Exclusion Criteria:

* Patients who are already enrolled in the study
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-08-09 (Actual); Primary Completion 2018-02-13 (Actual); Study Completion 2018-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Wyss, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Teaching Method A | Teaching Method B
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Teaching Method A | Teaching Method B | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (8) | 69 (13) | 70 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 9 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24
Average pain [Mean (Standard Deviation); unit: units on a 0-10 scale] — Average pain was assessed using a 0-10 scale, where 0 represents no pain and 10 represents worst possible pain. Higher scores represent worse outcomes.
  units on a 0-10 scale | 5.6 (2.2) | 4.8 (2.3) | 5.2 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Patient Satisfaction With the Teaching Method
Description: Satisfaction will be assessed using a 0-10 scale, where 0=not satisfied and 10=most satisfied. The higher the score, the greater the satisfaction.
Time Frame: 1 month post-injection
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teaching Method A | Teaching Method B
Number analyzed (Participants) | 12 | 12
units on a scale | 8.8 (1.6) | 8.3 (2.2)

2. Primary Outcome: Provider Satisfaction With the Teaching Method
Description: as for outcome 1
Time Frame: 1 month post-injection
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teaching Method A | Teaching Method B
Number analyzed (Participants) | 12 | 12
units on a scale | 6.0 (1.9) | 8.0 (1.0)

3. Primary Outcome: Patient Satisfaction With the Teaching Method
Description: as for outcome 1
Time Frame: 3 months post-injection
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teaching Method A | Teaching Method B
Number analyzed (Participants) | 12 | 12
units on a scale | 8.6 (2.2) | 8.6 (1.0)

4. Secondary Outcome: Number of Patients Who Would Have Preferred a Different Method of Receiving Education.
Description: Patient will be asked: "Would you have preferred a different method of receiving education?"
Time Frame: 3 months post-injection
Measure: Count of Participants; unit: Participants
Arm/Group | Teaching Method A | Teaching Method B
Number analyzed (Participants) | 12 | 12
Participants | 1 | 1

5. Secondary Outcome: Number of Patients Who Believed That the Education They Received Helped With the Care of Their Osteoarthritis
Description: Patient will be asked: "Did the education you received help with the care of your osteoarthritis?"
Time Frame: 3 months post-injection
Measure: Count of Participants; unit: Participants
Arm/Group | Teaching Method A | Teaching Method B
Number analyzed (Participants) | 12 | 12
Participants | 7 | 8

6. Secondary Outcome: PROMIS Physical Health Score
Description: The physical health score will be surveyed using the PROMIS-10 global health questionnaire. A higher score indicates better physical health. Scores range from 16.2 to 67.7.
Time Frame: 3 months post-injection
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Teaching Method A | Teaching Method B
Number analyzed (Participants) | 12 | 12
score on a scale | 45.8 (5.1) | 48.4 (6.5)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 3 months.
Arm/Group | Teaching Method A | Teaching Method B
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-25): https://cdn.clinicaltrials.gov/large-docs/63/NCT03245463/Prot_SAP_000.pdf